CLINICAL TRIAL: NCT03913143
Title: Double-masked, Randomized, Controlled, Multiple-dose Study to Evaluate Efficacy, Safety, Tolerability and Syst. Exposure of QR-110 in Leber's Congenital Amaurosis (LCA) Due to c.2991+1655A>G Mutation (p.Cys998X) in the CEP290 Gene
Brief Title: A Study to Evaluate Efficacy, Safety, Tolerability and Exposure After a Repeat-dose of Sepofarsen (QR-110) in LCA10 (ILLUMINATE)
Acronym: ILLUMINATE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ProQR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PQ-110-003; 2018-003501-25 (EudraCT Number)
Record Dates: First submitted 2019-02-21; First posted 2019-04-12 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Vision Disorders; Sensation Disorders; Neurologic Manifestations; Eye Diseases; Eye Diseases, Hereditary; Eye Disorders Congenital; Retinal Disease
Keywords: LCA10; CEP290; p.Cys998X; c.2991+1655A>G; Leber's Congenital Amaurosis; Antisense oligonucleotide; RNA therapy; QR-110; sepofarsen
MeSH Terms: conditions — Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Vision Disorders; Sensation Disorders; Neurologic Manifestations; Eye Diseases; Eye Diseases, Hereditary; Eye Abnormalities; Retinal Diseases; Meckel Syndrome, Type 4; Optic Atrophy, Hereditary, Leber | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Dose 1 sepofarsen (QR-110) (Experimental): Initial loading dose, followed by maintenance doses at month 3 and every 6 months there after, administered by intravitreal injection (24 months duration of treatment). After 12 months treatment of the contralateral eye may be initiated
  Interventions: Drug: sepofarsen
- Group 2: Dose 2 sepofarsen (QR-110) (Active Comparator): Initial loading dose, followed by maintenance doses at month 3 and every 6 months there after, administered by intravitreal injection (24 months duration of treatment). After 12 months treatment of the contralateral eye may be initiated
  Interventions: Drug: sepofarsen
- Group 3: Sham (Sham Comparator): Sham procedure (no experimental drug administered), Day 1, month 3 and every six months there after. After 12 months cross over to active study drug may be initiated
  Interventions: Other: Sham

INTERVENTIONS:
Drug: sepofarsen — RNA antisense oligonucleotide for intravitreal injection
  Other Names: QR-110
  Arms: Group 1: Dose 1 sepofarsen (QR-110); Group 2: Dose 2 sepofarsen (QR-110)
Other: Sham — Sham-Procedure (no experimental drug administered)
  Arms: Group 3: Sham

SUMMARY:
The purpose of this double-masked, randomized, controlled, multiple-dose study is to evaluate the efficacy, safety, tolerability and systemic exposure of sepofarsen (QR-110) administered via intravitreal injection in subjects with Leber's Congenital Amaurosis (LCA) due to the CEP290 p.Cys998X mutation after 24 months of treatment

DETAILED DESCRIPTION:
The purpose of this double-masked, randomized, controlled, multiple-dose study is to evaluate the efficacy, safety, tolerability and systemic exposure of sepofarsen (QR-110) administered via intravitreal injection in subjects with Leber's Congenital Amaurosis (LCA) due to the CEP290 p.Cys998X mutation after 24 months of treatment.

At study start subjects will be randomized to one of 3 treatment groups with either active study drug or sham treatment.

Sepofarsen (QR-110) will be administered via intravitreal (IVT) injection into the subject's treatment eye (the subject's worse eye).

Subjects in the sham-procedure group will undergo a procedure that will closely mimic the active injection.

After each dosing subjects will be assessed for safety and tolerability at follow up visits.

After the first eye has been treated for at least 12 months, treatment of the contralateral eye and cross-over of subjects assigned to sham procedure may be initiated in eligible eyes (in a masked manner) based on assessment of benefit/risk (including review of data from all clinical trials), and with concurrence of the Medical Monitor.

ELIGIBILITY:
Main Inclusion Criteria Relating to Study Initiation:

* Male or female, ≥ 8 years of age at Screening with a clinical diagnosis of LCA10 and a molecular diagnosis of homozygosity or compound heterozygosity for the c.2991+1655A>G mutation, based on genotyping analysis at Screening. A historic genotyping report from a certified laboratory is acceptable with Sponsor approval.
* BCVA better or equal to Logarithm of the Minimum Angle of Resolution (LogMAR) +3.0 (Hand Motion), and equal to or worse than LogMAR +0.4 in the treatment eye.
* Detectable outer nuclear layer (ONL) in the area of the macula.
* An electroretinogram (ERG) result consistent with LCA. A historic ERG result may be acceptable for eligibility.

Main Exclusion Criteria Relating to Study Initiation:

* Presence of any significant ocular or non-ocular disease/disorder (including medication and laboratory test abnormalities).
* Prior receipt of intraocular surgery, periocular surgery, or IVT injection within 1 month prior to study start or planned intraocular surgery or procedure during the course of the study.Subjects who received an intraocular or periocular surgery between 1 to 3 months prior Screening, may only be considered for inclusion if there are no clinically significant complications of surgery present, and following approval by the Medical Monitor.
* History or presence of ocular herpetic diseases.
* Presence of any active ocular infection in the either eye.
* Presence of lens opacities/cataracts in the treatment eye.
* Current treatment or treatment within the past 12 months with therapies known to influence the immune system.
* History of glaucoma, or an IOP greater than 24 mmHg, at is not controlled with medication.
* History of amblyopia
* Use of any investigational drug or device within 90 days or 5 half-lives of Day 1, whichever is longer, or plans to participate in another study of a drug or device during the PQ-110-003 study period.
* Any prior receipt of genetic or stem-cell therapy.
* Known hypersensitivity to antisense oligonucleotides or any constituents of the injection.
* Pregnant and breastfeeding subjects.

Main Inclusion Criteria Relating to Treatment Initiation Contralateral Eye:

* BCVA equal to or better than LP (logMAR +4), using the best BCVA reading at Month 12 and based on ETDRS or BRVT.
* Detectable outer nuclear layer (ONL) in the area of the macula.
* Clear ocular media and adequate pupillary dilation to permit good quality retinal imaging.

Main Exclusion Criteria Relating to Treatment Initiation Contralateral Eye:

* Presence of any significant ocular or non-ocular disease/disorder (including medication and laboratory test abnormalities).
* History or presence of ocular herpetic diseases.
* Presence of any active ocular infection in either eye.
* Presence of any lens opacities which are clinically significant, would adequately prevent clinical and photographic evaluation of the retina.
* A planned IVT injection or intraocular or periocular surgery/procedure (including refractive surgery) during the course of the study.
* A history of glaucoma or an IOP greater than 24 mmHg that is not controlled with medication.
* History of amblyopia.
* Plans to participate in another study of a drug or device during the study period.
* Pregnant and breastfeeding subjects.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in BCVA | 12 months
  Change in Best-corrected visual acuity (BCVA) relative to baseline after 12 months of treatment versus sham-procedure

SECONDARY OUTCOMES:
Change from baseline in BCVA ≤ -0.3 LogMAR | 12 and 24 months
  Change from baseline in BCVA in subjects with BCVA better than 1.7 Logarithm of the minimum angle of resolution (LogMAR) at baseline
Clinical meaningful improvement in subjects with BCVA ≤ 1.7 LogMAR | 12 and 24 months
  Change from baseline in BCVA by a clinically meaningful improvement in subjects with BCVA equal to or worse than 1.7 LogMAR at baseline.
Change in BCVA based on FrACT | 12 and 24 months
  Change from baseline in BCVA based on Freiburg visual acuity and contrast test (FrACT)
Change in mobility course score | 12 and 24 months
  Change from baseline in mobility course score
Change in ellipsoid zone (EZ) width/area assessed by SD-OCT | 12 and 24 months
  Change from baseline in ellipsoid zone (EZ) width/area assessed by SD-OCT
Change in oculomotor instability (OCI) | 12 and 24 months
  Change in oculomotor instability from baseline
Change in FST light sensitivity | 12 and 24 months
  Change from baseline in light sensitivity Full-field light sensitivity threshold (FST) testing (white, red, blue)
Change in LLVA | 12 and 24 months
  Change from baseline in low luminance visual acuity (LLVA)
Change in patient reported visual function via VFQ-25 (adults) | 12 and 24 months
  Change in patient reported visual function, as measured by the Visual Function Questionnaire-25 (VFQ-25) score for adult subjects relative to baseline
Change in patient reported visual function via CVAQC (pediatrics) | 12 and 24 months
  Change in patient reported visual function, as measured by the Cardiff Visual Ability Questionnaire for Children (CVAQC) for pediatric subjects relative to baseline
Change in the Patient Global Impressions of Severity (PGI-S) | 12 and 24 months
  Change in the patient-reported outcome (PRO) Patient Global Impressions of Severity (PGI-S)
Change in the Patient Global Impressions of Change (PGI-C) | 12 and 24 months
  Change in the PRO Patient Global Impressions of Change (PGI-C)
Change in FAF | 12 and 24 months
  Change from baseline as determined by fundus autofluorescence (FAF) imaging
Changes in microperimetry | 12 and 24 months
  Change from baseline as determined by microperimetry
Systemic exposure to QR-110 | 12 and 24 months
  Systemic exposure to QR-110
Ocular and non-ocular AEs | 12 and 24 months
  Frequency and severity of ocular and non-ocular AEs

CONTACTS AND LOCATIONS:
Overall Officials: ProQR Medical Monitor, Study Director — ProQR Therapeutics
Locations (14):
- University of Iowa, Iowa City, Iowa, United States
- Universitair Ziekenhuis Gent (UZ), Ghent, Belgium
- Brazil (2):
  - INRET Clínica/ Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Federal University of São Paulo - Hospital São Paulo (UNIFESP-HSP), São Paulo, São Paulo
- Canada (2):
  - The Hospital for Sick Children - SickKids, Toronto, Ontario
  - McGill University Health Centre - Centre for Innovative Medicine, Montreal, Quebec
- France (2):
  - Centre de maladies rares CHNO des Quinze Vingt, Paris
  - Hospital Civil de Strasbourg, Strasbourg
- Germany (2):
  - Justus-Liebig Universität - Department of Ophthalmology, Giessen
  - University of Tuebingen - Inst. for Ophthalmic Research, Tübingen
- Eye Clinic University of Campania Luigi Vanvitelli, Naples, Italy
- Netherlands (2):
  - Amsterdam University Medica Center - Locatie AMC, Amsterdam
  - Het Oogziekenhuis Rotterdam, Rotterdam
- Moorfields Eye Hospital - NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.proqr.com